CLINICAL TRIAL: NCT02940249
Title: Dose-response Effect of an Apple Extract on Postprandial Glycaemia: a Randomised Controlled Trial. The GLU-POMME Study.
Brief Title: Effects of an Apple Extract on Glycaemia: The GLU-Pomme Study
Acronym: GLU-Pomme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: DIANA Food (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: GLU-Pomme
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2018-03

CONDITIONS: Prevention of Hyperglycaemia
Keywords: Polyphenol; Apple; Fruit; Hyperglycaemia; Metabolic
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.2 g apple polyphenols (Experimental): 1200 mg apple polyphenols delivered in a low sugar drink.
  Interventions: Dietary Supplement: Apple polyphenols
- 0.9 g apple polyphenols (Experimental): 900 mg apple polyphenols delivered in a low sugar drink.
  Interventions: Dietary Supplement: Apple polyphenols
- 0.6 g apple polyphenols (Experimental): 600 mg apple polyphenols delivered in a low sugar drink.
  Interventions: Dietary Supplement: Apple polyphenols
- Placebo (Placebo Comparator): No polyphenols delivered in a low sugar drink.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Apple polyphenols — Drinks will be delivered in random order at 4 separate study visits immediately before a high-carbohydrate meal. Seven days wash-out period will be required between study days.
  Arms: 0.6 g apple polyphenols; 0.9 g apple polyphenols; 1.2 g apple polyphenols
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Postprandial hyperglycaemia can lead to adverse modifications to functional proteins within the body and eventually lead to the development of type 2 diabetes. Previous research by this group has shown that an apple polyphenol extract reduced hyperglycaemia following a high-carbohydrate meal. The aim of this study is to investigate the effects of lower doses of the apple extract on postprandial glycaemia, insulinaemia and plasma gastric inhibitory polypeptide concentrations following a mixed carbohydrate test meal.

DETAILED DESCRIPTION:
Introduction:

Sharp peaks in blood glucose levels can lead to adverse modifications to functional proteins, oxidative stress and pancreatic beta cell dysfunction. It is therefore desirable to consume a diet that will allow more gradual rises in blood glucose levels after meals. Fruit polyphenols may help to limit the glucose excursion following a high carbohydrate meal. Previous research by this research group has demonstrated that 1200 mg of apple polyphenols (Appl'In™) inhibited the average incremental area under the curve (T+0 to T+30 min) of plasma glucose by 54% relative to placebo. Possible mechanisms include inhibition of intestinal enzymes and inhibition of intestinal glucose absorption by decreasing SGLT1/GLUT2 transport activity. The literature also suggests that foods rich in polyphenols exert beneficial effects on risk factors of cardiovascular disease such as hypertension, lipid metabolism and vascular function.

Study design:

A randomised, controlled, double-blind, cross-over study will be conducted. Four matched test drinks will be consumed in random order on separate study visits immediately before a mixed-carbohydrate test meal, containing either: 1) 1.2 g, 2) 0.9 g 3). 0.6 g of apple polyphenols, or 4). placebo. Postprandial changes in plasma glucose, insulin, NEFA, GIP, GLP-1 concentrations as well as changes in vascular function will be measured. Twenty-four hour urine samples will be collected for analysis of urinary polyphenol metabolites and glucose. In a sub sample of participants, a paracetamol absorption test will be incorporated via addition of 1.5 g paracetamol into the test drink.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 y
* Male and female
* Healthy (free of diagnosed diseases listed in the exclusion criteria)
* Body Mass Index 18-35 kg/m2
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed written consent

Exclusion Criteria:

* Those diagnosed with Phenylketonuria (PKU)
* Those with known or suspected food and/or paracetamol intolerances, allergies or hypersensitivity
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are breast feeding
* Participation in another clinical trial
* Those who have donated blood within 3 months of the screening visit and participants for whom participation in this study would result in having donated more than 1500 millilitres of blood in the previous 12 months.
* Full Blood Counts and Liver Function test results outside of the normal range.
* Current smokers, or reported giving up smoking within the last 6 months
* History of substance abuse or alcoholism
* Reported history of Cardiovascular disease, diabetes (or fasting glucose ≥ 7.1 mmol/L), cancer, kidney, liver or bowel disease, gastrointestinal disorder or use of drug likely to alter gastrointestinal function
* Unwilling to restrict consumption of specified high polyphenol foods for 48 h before the study
* Weight change >3kg in preceding 2 months and body mass index <18 or >35 kg/m2
* Blood pressure ≥160/100 mmHg
* Total cholesterol ≥ 7.5 mmol/L; fasting triacylglycerol concentrations ≥ 5.0 mmol/L
* Medications that may interfere with the study: alpha-glucosidase inhibitors (acarbose: Glucobay), insulin sensitizing drugs (metformin: Glucophage, Glucophage SR, Eucreas, Janumet; thiazolidinediones: Actos, Competact), sulfonylureas (Daonil, Diamicron, Diamicron MR, Glibenese, Minodiab, Amaryl Tolbutamide), and lipid lowering drugs (statins, nicotinic acid, colestyramine anhydrous, ezetimibe, fibrates); and medications that may react unpredictably with paracetamol: ketoconazole, metoclopramide, carbamazepine, phenobarbital, phenytoin, primidone, warfarin and other products containing paracetamol. Other medications should be reviewed by medical representative from KCL on a case by case basis.
* Nutritional supplements that may interfere with the study: higher dose vitamins/minerals (>200% Recommend Nutrient Intake), B vitamins, Vitamin C, calcium, copper, chromium, iodine, iron, magnesium, manganese, phosphorus, potassium and zinc. Subjects already taking vitamin or minerals at a dose around 100% or less up to 200% of the RNI, or evening primrose/algal/fish oil supplements will be asked to maintain habitual intake patterns, ensuring that they take them every day and not sporadically. They will be advised not to stop taking supplements or start taking new supplements during the course of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01; Primary Completion 2017-11 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolic Research Unit at King's College London, Waterloo Campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants were recruited from King's College London (KCL) and the general public in London and surrounding counties.
Pre-assignment Details: 34 out of 64 screened were randomized. Of those not randomized, 8 did not meet inclusion criteria, 1 had a minor adverse event, and 21 declined to participate.
Groups:
- Doses of Apple Extract: Randomised sequences of singled doses of 0, 0.9, 1.2 and 1.8 g apple extract consumed with a test meal. Participants first received intervention 1 on the morning of a study visit, followed by a washout period of at least 7 days, then intervention 2 followed by a 7 day washout period, then intervention 3 followed by a 7 day washout period, then intervention 4.
Period: Overall Study
Arm/Group | Doses of Apple Extract
Started | 34
Completed | 30
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants completing all study interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Customized [Mean (Standard Deviation); unit: years] — Mean (SD) age (years) Population: Numbers analyzed in rows differ from overall as they are given for men, postmenopausal women, and premenopausal women separately.
  years
    Males: number analyzed (Participants) | 11
    Males | 30 (12)
    Premenopausal females: number analyzed (Participants) | 13
    Premenopausal females | 27 (8)
    Postmenopausal females: number analyzed (Participants) | 6
    Postmenopausal females | 56 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] — Fasting plasma glucose concentrations (mmol/L)
  mmol/L | 5.18 (0.39)

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glycaemia
Description: Primary outcome: Area over baseline t+0-30 min for plasma glucose
Time Frame: 30 min following the test drink
Measure: Mean (Standard Error); unit: mmol/L*min
Groups:
- 1.8 g Apple Extract: High dose of polyphenol apple extract in a drink
- 1.2 g Apple Extract: Medium dose of polyphenol apple extract in a drink
- 0.9 g Apple Extract: Low dose of apple extract in a drink
- 0 g Apple Extract: Control in a drink matched for appearance and macronutrients
Arm/Group | 1.8 g Apple Extract | 1.2 g Apple Extract | 0.9 g Apple Extract | 0 g Apple Extract
Number analyzed (Participants) | 30 | 30 | 30 | 30
mmol/L*min | 11.3 (1.2) | 15.2 (1.5) | 17.8 (1.6) | 27.1 (2.5)

2. Secondary Outcome: Postprandial Insulinaemia
Description: Peak postprandial insulin concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min.
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

3. Secondary Outcome: Postprandial Glucose-dependent Insulinotropic Polypeptide (GIP) Concentrations
Description: Peak postprandial GIP concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min.
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

4. Secondary Outcome: Postprandial Glucagon-like Peptide-1 (GLP-1) Concentrations
Description: Peak postprandial GLP-1 concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min.
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

5. Secondary Outcome: Postprandial C-peptide Concentrations
Description: Peak postprandial C-peptide concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min.
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

6. Secondary Outcome: Postprandial Non-esterified Fatty Acid (NEFA) Concentrations
Description: Peak postprandial NEFA concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

7. Secondary Outcome: Postprandial Triglyceride (TAG) Concentrations
Description: Peak postprandial TAG concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min.
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

8. Secondary Outcome: Postprandial Paracetamol Concentrations
Description: Peak postprandial paracetamol concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min (1.5 g paracetamol will be added to all test drinks in a sub-group of participants).
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

9. Secondary Outcome: Postprandial Polyphenol Metabolite Concentrations
Description: Peak postprandial polyphenol metabolites concentrations (Cmax) t +0-30 min and change from baseline data and areas over baseline t+0-30 min and t+0-240 min.
Time Frame: baseline and 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240 min following the test drink
Reporting Status: Not Posted

10. Secondary Outcome: Vascular Endothelial Function by Flow-mediated Dilation (FMD)
Description: Change in FMD after the consumption of test drink.
Time Frame: baseline and 120, 240, 300 min following the test drink
Reporting Status: Not Posted

11. Secondary Outcome: Vascular Function (Arteriograph Measurement)
Description: Change in augmentation index following the test drink.
Time Frame: Baseline and 60, 90, 120, 180, 240 min following the test drink
Reporting Status: Not Posted

12. Secondary Outcome: Blood Pressure
Description: Change in blood pressure following the test drink.
Time Frame: Baseline and 60, 90, 120, 180, 240 min following the test drink
Reporting Status: Not Posted

13. Secondary Outcome: Urinary Polyphenol Metabolites
Description: Change in urinary polyphenol metabolite concentration following the test drink.
Time Frame: 0-4 h, 4-8 h, 8-24 h following the test drink
Reporting Status: Not Posted

14. Secondary Outcome: Urinary Glucose
Description: Change in urinary glucose concentration following the test drink.
Time Frame: 0-4 h, 4-8 h, 8-24 h following the test drink
Reporting Status: Not Posted

15. Other Pre Specified Outcome: 7-day Food Diary
Description: Habitual dietary intake analysis
Time Frame: Baseline
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Women's Health Questionnaire
Description: Questionnaire to identify menstrual phase
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 hour study visit for each of the 4 interventions.
Description: Arms/groups for randomised sequence are combined as there are a large number of different sequences.
  All-Cause Mortality was not monitored/assessed.
Arm/Group | 1.8 g Apple Extract | 1.2 g Apple Extract | 0.9 g Apple Extract | 0 g Apple Extract
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02940249/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT02940249/ICF_001.pdf